CLINICAL TRIAL: NCT00629122
Title: Pharmacokinetic Evaluation of Sublingual Versus Oral Tacrolimus Administration in Patients Awaiting Kidney Transplantation
Brief Title: Pharmacokinetics of Sublingual Versus Oral Tacrolimus in Patients Awaiting Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 0710009492
Record Dates: First submitted 2008-02-12; First posted 2008-03-05 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Kidney Failure, Chronic
Keywords: Kidney Transplantation; Tacrolimus (Prograf); Pharmacokinetics; Sublingual administration; Drug interactions (Cytochrome P450 and p-glycoprotein)
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus; Clotrimazole; Deglutition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Tacrolimus and Nystatin Suspension (Experimental): Administer sublingual tacrolimus 2 mg every 12 hours (subject weight < 90 kg) or 3 mg every 12 hours (subject weight > 90kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth.
  Nystatin suspension 5 mL every 12 hours (study days 1 - 3 and 6 - 8).
  Interventions: Drug: Tacrolimus (Arm A); Drug: Nystatin Suspension
- B: Tacrolimus and Clotrimazole Troche (Experimental): Administer sublingual tacrolimus 1 mg every 12 hours (subject weight < 90 kg) or 2 mg every 12 hours (subject weight > 90 kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth.
  Clotrimazole troche 10 mg every 12 hours (study day 1 - 3 and 6 - 8).
  Interventions: Drug: Tacrolimus (Arm B); Drug: Clotrimazole Troche

INTERVENTIONS:
Drug: Tacrolimus (Arm B) — Study day 1 (9a): Initiate sublingual (SL) tacrolimus and clotrimazole troche x 5 doses; Study day 3 (9a): Collection of pharmacokinetic parameters around the 5th SL tacrolimus dose; Study day 3 (9p): Start washout period, no drug administration (tacrolimus, clotrimazole); Study day 5 (9p): End washout period; Study day 6 (9a): Initiate oral tacrolimus and clotrimazole troche x 5 doses; Study day 8 (9a): Collection of pharmacokinetic parameters around the 5th oral tacrolimus dose; Study day 15: Contact subject by telephone to assess for any adverse effects. To ensure that dietary intake does not affect the absorption profile of tacrolimus we will ensure that breakfast is given 15 minutes prior to drug administration on the days of pharmacokinetic assessment (study day 3 and 8).
  Other Names: Prograf
  Arms: B: Tacrolimus and Clotrimazole Troche
Drug: Clotrimazole Troche — Study day 1 (9a): Initiate sublingual (SL) tacrolimus and clotrimazole troche x 5 doses; Study day 3 (9a): Collection of pharmacokinetic parameters around the 5th SL tacrolimus dose; Study day 3 (9p): Start washout period, no drug administration (tacrolimus, clotrimazole); Study day 5 (9p): End washout period; Study day 6 (9a): Initiate oral tacrolimus and clotrimazole troche x 5 doses; Study day 8 (9a): Collection of pharmacokinetic parameters around the 5th oral tacrolimus dose; Study day 15: Contact subject by telephone to assess for any adverse effects. To ensure that dietary intake does not affect the absorption profile of tacrolimus we will ensure that breakfast is given 15 minutes prior to drug administration on the days of pharmacokinetic assessment (study day 3 and 8).
  Other Names: Mycelex
  Arms: B: Tacrolimus and Clotrimazole Troche
Drug: Tacrolimus (Arm A) — Study day 1 (9a): Initiate sublingual (SL) tacrolimus and nystatin suspension x 5 doses; Study day 3 (9a): Collection of pharmacokinetic parameters around the 5th SL tacrolimus dose; Study day 3 (9p): Start washout period, no drug administration (tacrolimus, nystatin); Study day 5 (9p): End washout period; Study day 6 (9a): Initiate oral tacrolimus and nystatin suspension x 5 doses; Study day 8 (9a): Collection of pharmacokinetic parameters around the 5th oral tacrolimus dose; Study day 15: Contact subjects by telephone to assess for any adverse effects. To ensure that dietary intake does not affect the absorption profile of tacrolimus we will ensure that breakfast is given 15 minutes prior to drug administration on the days of pharmacokinetic assessment (study day 3 and 8).
  Other Names: Prograf
  Arms: A: Tacrolimus and Nystatin Suspension
Drug: Nystatin Suspension — Study day 1 (9a): Initiate sublingual (SL) tacrolimus and nystatin suspension x 5 doses; Study day 3 (9a): Collection of pharmacokinetic parameters around the 5th SL tacrolimus dose; Study day 3 (9p): Start washout period, no drug administration (tacrolimus, nystatin); Study day 5 (9p): End washout period; Study day 6 (9a): Initiate oral tacrolimus and nystatin suspension x 5 doses; Study day 8 (9a): Collection of pharmacokinetic parameters around the 5th oral tacrolimus dose; Study day 15: Contact subjects by telephone to assess for any adverse effects. To ensure that dietary intake does not affect the absorption profile of tacrolimus we will ensure that breakfast is given 15 minutes prior to drug administration on the days of pharmacokinetic assessment (study day 3 and 8).
  Other Names: Nystatin Swish and Swallow
  Arms: A: Tacrolimus and Nystatin Suspension

SUMMARY:
Tacrolimus (Prograf) belongs to a class of medications known as the calcineurin inhibitors. It is a maintenance drug that is used to prevent rejection in kidney, liver, and heart transplant recipients. Calcineurin inhibitors display high pharmacokinetic (the body's effects on a drug) variability and necessitate use of blood tests to ensure that adequate drug levels are present to maintain effectiveness and safety. Early after transplant or at times when tacrolimus cannot be taken by mouth, alternative routes of administration are sought. Although an intravenous (through the vein) product is available, it can be toxic to the kidneys and has been associated with allergic reactions. Drug delivery via the oral mucosa is an alternative method of systemic drug administration which offers an alternative when oral administration is impractical (gastrointestinal dysmotility, reduced drug absorption, intestinal failure, difficulty in swallowing, or in those with nausea or vomiting). Administration of tacrolimus by the sublingual route may allow for direct entry into the systemic circulation and bypasses problems associated with drug absorption and breakdown that take place in the small intestine.

DETAILED DESCRIPTION:
Tacrolimus (Prograf) belongs to a class of medications known as the calcineurin inhibitors. It is a maintenance drug that is used to prevent rejection in kidney, liver, and heart transplant recipients. Calcineurin inhibitors display high pharmacokinetic (the body's effects on a drug) variability and necessitate use of blood tests to ensure that adequate drug levels are present to maintain effectiveness and safety. The amount of oral tacrolimus that is absorbed varies in all patient populations studied. Tacrolimus is metabolized or broken down for elimination by the liver and small intestine via cytochrome P450 (CYP)3A4, CYP 3A5, and p-glycoprotein enzyme systems. Enzyme activity is affected by several single nucleotide polymorphisms (SNPs) in an individuals genetic make-up and differences in expression may contribute to variations in tacrolimus pharmacokinetics. There are number of drug-drug interactions where concomitantly administered medications can increase or decrease this break down of tacrolimus. Early after transplant or at times when tacrolimus cannot be taken by mouth, alternative routes of administration are sought. Although an intravenous (through the vein) product is available, it can be toxic to the kidneys and has been associated with allergic reactions. Studies in lung transplant recipients have utilized sublingual (under the tongue) tacrolimus administration with successful outcomes. Drug delivery via the oral mucosa is an alternative method of systemic drug administration which offers an alternative when oral administration is impractical (gastrointestinal dysmotility, reduced drug absorption, intestinal failure, difficulty in swallowing, or in those with nausea or vomiting). Administration of tacrolimus by the sublingual route allows for direct entry into the systemic circulation and bypasses problems associated with drug absorption and breakdown that take place in the small intestine. In order to learn more about the possible role of sublingual tacrolimus among transplant recipients we will administer tacrolimus sublingually. In addition, we will evaluate differences in expression and bioactivity of SNP polymorphisms and their effects in tacrolimus pharmacokinetics. Patients awaiting kidney transplantation who are listed on the kidney transplant waiting list or those with upcoming living donor transplants at our center will be administered five doses of sublingual tacrolimus followed by five doses of oral tacrolimus. We will evaluate and then compare the pharmacokinetic characteristics of sublingual and oral tacrolimus administration among the study participants. The purpose of this study is to assess the pharmacokinetic and pharmacodynamic parameters of tacrolimus after sublingual and oral administration. A secondary objective is to assess the drug-drug interaction between concomitant therapy with clotrimazole.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients awaiting kidney transplantation aged ≥ 18 years

Exclusion Criteria:

* Patients concurrently treated with medications that interact with tacrolimus (other than clotrimazole)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith J Aull, Pharm.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NewYork-Presbyterian Hospital, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Tacrolimus and Nystatin): Sublingual (SL) tacrolimus 2 mg every 12 hours (subject weight < 90 kg) or 3 mg every 12 hours (subject weight > 90kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral (PO) tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth. Nystatin suspension 5 mL every 12 hours (study days 1 - 3 and 6 - 8).
  Study day 1: Initiate SL tacrolimus and nystatin suspension x 5 doses. Study day 3: Collection of pharmacokinetic parameters around 5th SL tacrolimus dose.
  Study day 3: Start washout period, no drug administration (tacrolimus, nystatin).
  Study day 5: End washout period. Study day 6: Initiate PO tacrolimus and nystatin suspension x 5 doses. Study day 8: Collection of pharmacokinetic parameters around the 5th PO tacrolimus dose.
  Study day 15: Participants will be contacted by telephone to assess for any adverse effects.
- Arm B (Tacrolimus and Clotrimazole): Sublingual (SL) tacrolimus 1 mg every 12 hours (subject weight < 90 kg) or 2 mg every 12 hours (subject weight > 90 kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral (PO) tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth. Clotrimazole troche 10 mg every 12 hours (study day 1 - 3 and 6 - 8).
  Study day 1: Initiate SL tacrolimus and clotrimazole troche x 5 doses. Study day 3: Collection of pharmacokinetic parameters around the 5th SL tacrolimus dose.
  Study day 3: Start washout period, no drug administration (tacrolimus, clotrimazole).
  Study day 5: End washout period.
  Study day 6: Initiate PO tacrolimus and clotrimazole troche x 5 doses. Study day 8: Collection of pharmacokinetic parameters around the 5th PO tacrolimus dose.
  Study day 15: Participants will be contacted by telephone to assess for any adverse effects.
Period: First Period: Day 1- 3 (Sublingual)
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole)
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0
Period: Second Period: Day 3-5 (Washout)
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole)
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0
Period: Third Period: Day 6-8 (Oral)
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole)
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A (Tacrolimus and Nystatin): Sublingual (SL) tacrolimus 2 mg every 12 hours (subject weight < 90 kg) or 3 mg every 12 hours (subject weight > 90kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral (PO) tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth. Nystatin suspension 5 mL every 12 hours (study days 1 - 3 and 6 - 8).
- Arm B (Tacrolimus and Clotrimazole): Sublingual (SL) tacrolimus 1 mg every 12 hours (subject weight < 90 kg) or 2 mg every 12 hours (subject weight > 90 kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral (PO) tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth. Clotrimazole troche 10 mg every 12 hours (study day 1 - 3 and 6 - 8).
- Total: Total of all reporting groups
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole) | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: C0 (ng/mL)
Description: Trough concentration
Time Frame: Day 3 and Day 8, time 0 (before tacrolimus dose)
Measure: Median (Full Range); unit: ng/mL
Groups:
- Arm A (Tacrolimus and Nystatin): Sublingual tacrolimus 2 mg every 12 hours (subject weight < 90 kg) or 3 mg every 12 hours (subject weight > 90kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth. Nystatin suspension 5 mL every 12 hours (study days 1 - 3 and 6 - 8).
- Arm B (Tacrolimus and Clotrimazole): Sublingual tacrolimus 1 mg every 12 hours (subject weight < 90 kg) or 2 mg every 12 hours (subject weight > 90 kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth. Clotrimazole troche 10 mg every 12 hours (study day 1 - 3 and 6 - 8).
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole)
Number analyzed (Participants) | 2 | 3
ng/mL
  Day 3 (Sublingual) | 1.45 [0.1 to 2.8] | 6.2 [3.0 to 8.3]
  Day 8 (Oral) | 1.25 [0.2 to 2.3] | 6.5 [3.2 to 11.2]

2. Primary Outcome: Cmax
Description: Maximum concentration (ng/mL)
Time Frame: Day 3 and Day 8, at time of maximum concentration
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole)
Number analyzed (Participants) | 2 | 3
ng/mL
  Day 3 (Sublingual) | 9.6 [2.0 to 17.2] | 14.0 [6.5 to 22.5]
  Day 8 (Oral) | 4.6 [3.2 to 6.0] | 19.5 [10.1 to 19.8]

3. Primary Outcome: Tmax
Description: Time to Maximum concentration (hours)
Time Frame: Day 3 and Day 8, time of maximum concentration
Measure: Median (Full Range); unit: hours
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole)
Number analyzed (Participants) | 2 | 3
hours
  Day 3 (Sublingual) | 1.75 [1.5 to 2.0] | 3.0 [1.5 to 4.0]
  Day 8 (Oral) | 0.875 [0.75 to 1.0] | 2.0 [2.0 to 4.0]

4. Primary Outcome: Estimated AUC 0-6
Description: Area Under the Concentration-Time Curve from 0-6 hours (mg-hr/L)
Time Frame: Day 3 and Day 8, calculated based on concentrations measured between hours 0 and 6
Measure: Number; unit: mg-hr/L
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole)
Number analyzed (Participants) | 2 | 3
mg-hr/L
  Patient 1 Sublingual (day 3) | 9.3 | NA — The patient did not receive that combination (ie. was in other arm)
  Patient 1 Oral (day 8) | 4.9 | NA — The patient did not receive that combination (ie. was in other arm)
  Patient 2 Sublingual (day 3) | NA — The patient did not receive that combination (ie. was in other arm) | 27.2
  Patient 2 Oral (day 8) | NA — The patient did not receive that combination (ie. was in other arm) | 32.4
  Patient 3 Sublingual (day 3) | NA — The patient did not receive that combination (ie. was in other arm) | 66.0
  Patient 3 Oral (day 8) | NA — The patient did not receive that combination (ie. was in other arm) | 76.0
  Patient 4 Sublingual (day 3) | NA — The patient did not receive that combination (ie. was in other arm) | 63.7
  Patient 4 Oral (day 8) | NA — The patient did not receive that combination (ie. was in other arm) | 52.5
  Patient 5 Sublingual (day 3) | 63.0 | NA — The patient did not receive that combination (ie. was in other arm)
  Patient 5 Oral (day 8) | 23.2 | NA — The patient did not receive that combination (ie. was in other arm)

5. Primary Outcome: Tacrolimus Powder Dissolution Time
Description: Tacrolimus Powder Dissolution Time during Sublingual Administration (minutes)
Time Frame: Day 3, minutes to powder dissolution
Measure: Median (Full Range); unit: minutes
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole)
Number analyzed (Participants) | 2 | 3
minutes | 2.25 [2.0 to 2.5] | 2.0 [1.5 to 3.0]

6. Secondary Outcome: Drug Interactions and Genotypes
Description: Impact of drug interaction between tacrolimus and clotrimazole troche vs. nystatin suspension. Evaluate genotype polymorphisms that influence CYP3A4, CYP3A5, and p-glycoprotein expression to determine impact on sublingual and oral tacrolimus delivery.
Time Frame: 2 weeks
Population: We were unable to assess genotype polymorphisms due to the small number of subjects enrolled in the study.
Arm/Group | Arm A (Tacrolimus and Nystatin) | Arm B (Tacrolimus and Clotrimazole)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Arm A (Tacrolimus + Nystatin): Sublingual tacrolimus 2 mg every 12 hours (subject weight < 90 kg) or 3 mg every 12 hours (subject weight > 90kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth. Nystatin suspension 5 mL every 12 hours (study days 1 - 3 and 6 - 8).
- Arm B (Tacrolimus + Clotrimazole): Sublingual tacrolimus 1 mg every 12 hours (subject weight < 90 kg) or 2 mg every 12 hours (subject weight > 90 kg) (study day 1 - 3). Tacrolimus capsules will be opened and the contents placed under the participants tongue. Oral tacrolimus at same dose every 12 hours (study day 6 - 8). Tacrolimus capsules will be administered by mouth. Clotrimazole troche 10 mg every 12 hours (study day 1 - 3 and 6 - 8).
Arm/Group | Arm A (Tacrolimus + Nystatin) | Arm B (Tacrolimus + Clotrimazole)
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Tacrolimus + Nystatin) (N=2) | Arm B (Tacrolimus + Clotrimazole) (N=3)
Bitter taste in mouth (Gastrointestinal disorders) | 2 (2) | 3 (3) — Bitter taste of the tacrolimus powder for sublingual administration.

LIMITATIONS AND CAVEATS:
Small sample size; variable absorption profile; poor vascular access in some subjects; possible enteral absorption of sublingual drug; unable to assess genotype polymorphisms due to the small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No